CLINICAL TRIAL: NCT01641419
Title: Randomized, Controlled Trial Comparing Duration of Analgesia After Popliteal Fossa Sciatiac Nerve Block With Ropivacaine 0.5% When Combined With Placebo, Dexamethasone 4mg or Dexamethasone 8 mg
Brief Title: Trial Comparing Duration of Analgesia After Popliteal Fossa Sciatiac Nerve Block With Ropivacaine 0.5% When Combined With Placebo, Dexamethasone 4mg or Dexamethasone 8 mg
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit subjects at our hospital due to change in surgical patient population. Not worth to continue.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jaime Ortiz, Assistant Professor of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-30398
Record Dates: First submitted 2012-07-11; First posted 2012-07-16 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Pain, Sciatic Block
Keywords: Pain; Ropivacaine; sciatic block; dexamethasone
MeSH Terms: conditions — Pain | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Ropivacaine 0.5% plus 2ml of normal saline used for nerve block
  Interventions: Drug: Placebo
- Dexamethasone 4 mg (Active Comparator): Ropivacaine 0.5% plus 2ml of dexamethasone 4 mg used for nerve block
  Interventions: Drug: Dexamethasone 4 mg
- Dexamethasone 8 mg (Active Comparator): Ropivacaine 0.5% plus 2ml of dexamethasone 8 mg used for nerve block
  Interventions: Drug: Dexamethasone 8 mg

INTERVENTIONS:
Drug: Placebo — 2 ml of saline added to 30 ml of ropivacaine 0.5% solution for nerve block
  Arms: Placebo
Drug: Dexamethasone 4 mg — 2 ml of dexamethasone 4 mg solution added to 30 ml of ropivacaine 0.5% solution for nerve block
  Arms: Dexamethasone 4 mg
Drug: Dexamethasone 8 mg — 2 ml of dexamethasone 8 mg solution added to 30 ml of ropivacaine 0.5% solution for nerve block
  Arms: Dexamethasone 8 mg

SUMMARY:
The purpose is to find out if the addition of dexamethasone to ropivacaine 0.5% increases the duration of pain relief provided by popliteal sciatic nerve block performed for foot/ankle surgery. The investigators also want to find out if there is a difference between 4 and 8 mg dose of dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-64
* ASA Physcial Status classification 1-3
* Foot and ankle surgery at Ben Taub General Hospital

Exclusion Criteria:

* diabetes mellitus
* peripheral neuropathy
* coagulopathy
* allergy to study drugs
* systemic glucocorticoid treatment (for 2 weeks or more) within 6 months of surgery
* chronic opioid use at home
* patient inability to properly describe pain to investigators
* pregancy
* prisoners
* patient or surgeon refusal

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | 48 hours
  Duration of analgesia of popliteal fossa sciatic nerve block defined as time of first pain as described by patient minus time of block placement in minutes

SECONDARY OUTCOMES:
Total pain medication | 24 hours
  Total amounts of morphine, fentanyl and hydrocodone/acetaminophen that the patient required for pain control during first 24 hours after surgery.
  All patients, regardless of group, will receive a standardized postoperative pain medication regimen which will include hydrocodone/acetaminophen tablets primarily, and morphine/fentanyl as needed.
Pain scores | 24 hours
  Pain score measured of numeric analog scale from 0-10 during first 24 hours measures and 0,1,2,4,8,12, and 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States